CLINICAL TRIAL: NCT05417854
Title: Ultrasound Treatment for Rheumatoid Arthritis Study [ULTRA Study]
Acronym: ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SecondWave Systems Inc. (Industry)
Collaborators: University of Minnesota (Other); DARPA (United States Department of Defense) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00062049; 140D0419C0092 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ultrasound Group (Experimental)
  Interventions: Device: Splenic Ultrasound

INTERVENTIONS:
Device: Splenic Ultrasound — Daily ultrasound application to the spleen of approximately 18 minutes per day, 5 days per week for up to 8 weeks, in addition to standard clinical care.
  Other Names: SecondWave Systems investigational MINI device

SUMMARY:
The research objective is to assess efficacy of spleen ultrasound stimulation in the treatment of rheumatoid arthritis (RA) in a pilot study.

Specific Aims:

* Measure RA disease activity and clinical metrics during and after an 8-week course of spleen-directed daily ultrasound treatments.
* Measure molecular correlates, including Erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), cortisol and cytokine levels, of rheumatoid arthritis disease activity during spleen-directed daily ultrasound treatments.

DETAILED DESCRIPTION:
Ultrasound is widely used in human medicine because it is safe, non-invasive, and painless. The same kind of ultrasound that is used for imaging (for example, to visualize babies in utero) may be able to treat inflammatory diseases including Rheumatoid Arthritis.

Multiple studies in animals with hyper-inflammation conditions (e.g., inflammatory arthritis and sepsis/lipopolysaccharide [LPS] injections) and recent human studies (e.g., for the treatment of joint inflammation in Rheumatoid Arthritis) have shown that ultrasound applied to the spleen can suppress blood/genetic markers of inflammation.

This study will employ investigational ultrasound devices produced by SecondWave Systems called the MINI ultrasound system.

This is a pilot single-arm treatment trial in which up to 15 study participants will receive noninvasive splenic-ultrasound therapy over eight weeks (five daily stimulation sessions per week). Clinical outcomes will be compared from baseline to end of the 8-week treatment period. Investigational splenic-ultrasound therapy will be delivered with the SecondWave MINI ultrasound system. The objective of the study is to assess the safety and potential efficacy for the MINI system for treatment of Rheumatoid Arthritis.

For ultrasound stimulation, a small wearable ultrasound device is positioned on the upper left abdomen area over the ribs. Study personnel will use an ultrasound imaging device to locate the spleen and to position the wearable MINI device in a proper location around the ribs area. Daily stimulation consists of an approximately 18-minute period for application of ultrasound to the spleen. Collection of clinical outcome data, patient-reported assessments, and blood draws collected at the 5 study visits to assess biomarkers of inflammation will be performed in each participant throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18 and above
2. Must carry a diagnosis of rheumatoid arthritis, as defined by the American College of Rheumatology in 2010: (https://www.rheumatology.org/Portals/0/Files/2010_revised_criteria_classification_ra.pdf)

   - Classification as "definite RA" is based on the confirmed presence of synovial thickening in at least 1 joint, absence of an alternative diagnosis that better explains the synovitis, and achievement of a total score of 6 or greater (of a possible 10) from the individual scores in 4 domains: number and site of involved joints (score range 0-5), serologic abnormality (score range 0-3), elevated acute-phase response (score range 0-1), and symptom duration (2 levels; range 0-1)
3. Exhibiting symptoms or signs of inadequate inflammatory disease control according to one of two measures:

   1. Multidimensional HAQ score of greater than 0.3
   2. DAS-28-CRP greater than 3.2 (http://www.phusewiki.org/wiki/index.php?title=Disease_Activity_Score_-_CRP_(DAS-CRP)
4. Candidate participant's rheumatoid arthritis medical therapy should be stable for two weeks leading up to the study. Moreover, participants must be willing to maintain their current medication regimen throughout the study enrollment period (in adjunct to the additional investigational ultrasound treatment)

Exclusion Criteria:

1. Active bacterial or viral infection
2. Pregnant women or those trying to become pregnant
3. Receiving active chemotherapy or immunotherapy to treat malignancy within 30 days prior to enrollment
4. Having received Rituximab monoclonal antibody medication within 30 days prior to enrollment
5. Presence of an implanted device
6. Asplenia
7. Splenomegaly
8. Ascites
9. Recent abdominal surgery
10. Currently participating in an investigational drug or device study
11. Open wound/sores near stimulation sites
12. Inability to perform minimal daily self-cares associated with feeding/dressing, according to HAQ
13. Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Within-arm change in the Disease Activity Score (DAS-28-CRP) from baseline to the completion of an up-to 8-week treatment period. | 8 weeks
  A decrease in Disease Activity Score indicates an improved outcome.

OTHER OUTCOMES:
Within-arm change of serum c-reactive protein (CRP) concentration. | 8 weeks
Within-arm change of serum erythrocyte sedimentation rate (ESR). | 8 weeks
Within-arm change of serum cortisol levels. | 8 weeks
Within-arm change of serum Tumor Necrosis Factor (TNFa) concentration. | 8 weeks
Within-arm change of serum Interleukin-1 beta (IL-1beta) concentration. | 8 weeks
Within-arm change of serum Interleukin-6 (IL-6) concentration. | 8 weeks
Within-arm change of serum Interleukin-6 (IL-8) concentration. | 8 weeks
Within-arm change of serum Interferon gamma (IFN-gamma) concentration. | 8 weeks
Within-arm change on the Multidimensional Health Assessment Questionnaire (HAQ). | 8 weeks
  A decreased score on the HAQ indicates an improved outcome.
Within-arm change on the EQ-5D health questionnaire. | 8 weeks
  A decreased score on questions from the EQ-5D indicates an improved outcome.
Exit interview questions. | End of study participation
  These questions ask the participant about whether they feel that they have benefited from the investigational treatment, whether they would recommend the investigational treatment to others, and the comfort level of the investigational treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Peterson, M.D., Principal Investigator — University of Minnesota Medical School, Division of Rheumatic and Autoimmune Diseases
Locations (2):
- United States (2):
  - University of Minnesota - Phillips-Wangensteen Building, Minneapolis, Minnesota
  - University of Minnesota Health Clinics and Surgery Center, Minneapolis, Minnesota